CLINICAL TRIAL: NCT00536900
Title: Abstinence-Linked Money Management
Brief Title: Clinical Trial of Abstinence-Linked Money Management
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0403026478; R01DA012952 (NIH)
Record Dates: First submitted 2007-09-26; First posted 2007-09-28 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2014-07

CONDITIONS: Substance Abuse
Keywords: Substance abuse; Behavior therapy; representative payee; cocaine abuse; alcohol abuse; case management; dual diagnosis
MeSH Terms: conditions — Substance-Related Disorders; Cocaine-Related Disorders; Alcoholism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Advisor-Teller Money Manager
  Interventions: Behavioral: Advisor-Teller Money Manager
- 2 (Active Comparator): FIT (finance instruction therapy)
  Interventions: Behavioral: FIT

INTERVENTIONS:
Behavioral: Advisor-Teller Money Manager — The acronym for the functions of ATM are TTT-- Teller (storing patient funds), Training patients by making and reviewing monthly budgets, and Treatment-Linked Spending in which weekly behavioral contracts link disbursement to completion of abstinence-related activities
  Arms: 1
Behavioral: FIT — FIT (finance instruction therapy) involves review of a financial workbook and budgeting sheets
  Arms: 2

SUMMARY:
This is a randomized controlled trial to test whether a money-management based intervention reduces substance abuse.

DETAILED DESCRIPTION:
While the Social Security Administration (SSA) no longer provides benefits for individuals disabled by drug abuse per se, approximately 50% of recipients have a concomitant substance abuse disorder. Supported by disability payments, this substance abuse impedes recovery/remission from the comorbid mental disorder. Money management is widely implemented in dual diagnosis treatment - in patients assigned payees to manage their funds and in patients receiving case management - but whether money management reduces substance abuse is unproven. If shown to be effective, money management-based therapy can be logically integrated into these existing arrangements. There is no specific substance abuse focus to standard payee and case management arrangements.

We have developed a money management-based therapy called Advisor-Teller money manager (the bank-like acronym is ATM). ATM involves having a patient voluntarily allow a therapist/money manager to limit the patients' access to his/her funds, thus preventing unrestricted access to cash from cueing substance use. Patients meet with therapist/money managers at least weekly. Meetings begin with a review of the previous week's expenditures, including expenditures for drugs and alcohol, and an on-site urine toxicology test and breathalyzer. Patients then plan a budget that is incompatible with drug use by budgeting funds for direct payment of expenses (such as rent), abstinence-compatible activities and long-term goals. Budgeting and planning will develop patients' skills at managing their funds. Dispensing procedures build upon the principles of therapeutic contracting. Patients contract to receive their funds for specific expenditures and then review the next week whether the funds were spent as planned.

We are conducting a Stage 2 randomized clinical trial in which 120 patients will be randomly assigned to 36-weeks of either ATM or Finance Instruction Therapy (FIT), a low intensity intervention in which patients are given basic financial instruction to determine the efficacy of ATM in reducing substance use.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older.
2. History of cocaine or alcohol abuse in the past 5 years
3. Global Assessment of Functioning score below 65.
4. Income of at least $450 per month.
5. Able to provide informed consent, as evidenced by being able to answer questions about the study (described in Human Subjects).
6. Enrolled at the New Haven Connecticut Mental Health Center (CMHC).
7. Able to provide at least 2 names, addresses and telephone numbers of at least 2 individuals who are likely to have knowledge of their whereabouts throughout study follow-up.

Exclusion Criteria:

1. Evidence of physiological dependence on sedatives or alcohol requiring a detoxification.
2. Has a conservator or a representative payee
3. Already receiving active money management (e.g. by case manager) in which the therapist/money manager makes more than one direct payment per month on behalf of the beneficiary.
4. Mentally Retarded, as evidenced by a DSM IV diagnosis of mental retardation or a clinical diagnosis of mental retardation.
5. Individuals in recovery from pathological gambling.
6. Individuals whose partner or spouse who co-manage their money is already enrolled in the study.
7. In the opinion of the Principal Investigator, the patient is unable to comply with the protocol procedures as evidenced by behavior or clinical information obtained during the enrollment and screening process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2004-06; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
weeks of abstinence | 36 weeks

SECONDARY OUTCOMES:
Dollars spent on alcohol | 36 weeks
Dollars spent on drugs | 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marc I Rosen, M.D., Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Rosen MI, Rounsaville BJ, Ablondi K, Black AC, Rosenheck RA. Advisor-Teller Money Manager (ATM) therapy for substance use disorders. Psychiatr Serv. 2010 Jul;61(7):707-13. doi: 10.1176/ps.2010.61.7.707. PMID 20592006